CLINICAL TRIAL: NCT06363305
Title: Impact of Sex in the Effect of Dietary Capsaicin on Cardiovascular Health: A Randomized Controlled Trial
Brief Title: Impact of Sex in the Effect of Dietary Capsaicin on Cardiovascular Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Skidmore College (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2402-1139
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Pre Hypertension; Hypertension
Keywords: vascular stiffness; blood pressure; vascular function
MeSH Terms: conditions — Prehypertension; Hypertension | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Parallel: Participants are randomly assigned to one of two groups in parallel for the duration of the study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The capsules will be placed into solid white color bottles, and labeled discreetly by a third party not directly involved with the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Capsaicin (Experimental): Over-the-counter dose of 2 x 440 mg capsules (880 mg, Capsicum Pepper Blend, Daily Manufacturing, Rockwell, North Carolina, USA)
  Interventions: Dietary Supplement: Dietary capsules
- Placebo (Placebo Comparator): The placebo will be 2 x 400-500 mg fiber (800 mg psyllium husk) capsules which were chosen to be of similar appearance (size, coloration, and texture).
  Interventions: Dietary Supplement: Dietary capsules

INTERVENTIONS:
Dietary Supplement: Dietary capsules — Daily doses of dietary capsaicin or placebo in capsule form

SUMMARY:
The investigators long-term goal is to better understand novel interventions to promote cardiovascular health in humans. The goal of the proposed research is to investigate whether there is sex-specificity in the effects of dietary capsaicin on mechanisms regulating nitric oxide (NO) bioavailability, its effect on key markers of cardiovascular (CV) health, including BP, macro- and microvascular function, and arterial stiffness. This knowledge will provide critical insight into the effects of dietary capsaicin on CV health and will guide future trials.

DETAILED DESCRIPTION:
Specific Aim 1: Determine the sex-specific effects of dietary capsaicin on central and peripheral blood pressure and arterial stiffness. The investigators hypothesize that dietary capsaicin intervention (6 week) will improve BP and arterial stiffness, likely in a sex-dependent manner. The investigators will measure heart rate variability and excretion of capsaicin and metabolites to ascertain bioavailability, and understand the mechanistic role of the autonomic nervous system, in capsaicin's effect on BP.

Specific Aim 2: Assess whether dietary capsaicin effects on vascular function is sex-specific. The investigators hypothesize that dietary capsaicin intervention (6 week) will improve NO bioavailability, through improved redox balance and lowered asymmetric dimethylarginine, thereby improving peripheral vascular function, likely in a sex-dependent manner.

Utilizing a double-blind, randomized, placebo-controlled, design the investigators will investigate whether there is sex-specificity in the effects of a 6-week dietary capsaicin intervention on nitric oxide (NO) bioavailability, BP, vascular function, and arterial stiffness.

ELIGIBILITY:
Inclusion Criteria:

* relatively healthy (other than elevated blood pressure) non-smoking men and women over the age of 18 from the local community

Exclusion Criteria:

* Women who are without a period (not due to a birth control method, intrauterine device or menopause), are pregnant, attempting to conceive, or are breastfeeding will be excluded.
* uncontrolled hypertension
* Anyone with severe illness or compromised or suppressed immune system (e.g. taking immune suppressants, chronic viral infection or treatment).
* Any participants with excessive sensitivity to spicy foods or fiber (psyllium husk) will be excluded
* Participants with food allergies will be excluded
* Participants who have difficulty swallowing or swallowing pills may be excluded.
* Participants who suffer from heartburn, hiatal hernia, gastritis, or peptic ulcer disease may be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure and Vascular Stiffness | Baseline, 24 hours, and 6-weeks
  The investigators will assess peripheral and estimated central blood pressures and vascular stiffness using pulse wave analysis.
Heart Rate (HR) and HR variability (HRV) | Baseline, 24 hours, and 6-weeks
  The investigators will assess HR and HRV using electrocardiogram and standard techniques to determine time and frequency domain estimates of HRV.
Flow Mediated Dilation | Baseline, 24 hours, and 6-weeks
  The investigators will assess brachial artery flow-mediated dilation using ischemia-reperfusion and ultrasound doppler to assess the dilatory capacity and reactive hyperemia.
Passive Leg Movement Hyperemia | Baseline, 24 hours, and 6-weeks
  The investigators will assess the hyperemic response to passive leg movement using ultrasound doppler.
Near Infrared Spectroscopy (NIRS) Vascular Occlusion Test | Baseline, 24 hours, and 6-weeks
  The investigators will assess the metabolic capacity and vascular reactivity using ischemia-reperfusion and NIRS

SECONDARY OUTCOMES:
Urinary Capsaicinoids | Baseline, 24 hours, and 6-weeks
  The investigators will collect urine to determine urinary capsaicin and associated metabolites to understand bioavailability and potential relation to function.
Blood Lipids | Baseline and 6-weeks
  The investigators will collect blood to determine blood lipids (cholesterol) and glucose.

CONTACTS AND LOCATIONS:
Locations (1):
- Skidmore College, Saratoga Springs, New York, United States

IPD SHARING:
Plan to Share IPD: No
Only deidentified data may be shared with the sponsor or research community through appropriate data repositories.